CLINICAL TRIAL: NCT00919763
Title: A Four-Week, Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of CD2027 Ointment 3 mcg/g Twice Daily in the Treatment of Adults With at Least Moderate Atopic Dermatitis
Brief Title: Efficacy and Safety Study of CD2027 Ointment 3 Microgram Per Gram (mcg/g) Twice Daily Treatment for Adults With at Least Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18158
Record Dates: First submitted 2009-06-09; First posted 2009-06-12 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-05

CONDITIONS: Atopic Dermatitis
Keywords: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD2027 Ointment 3 mcg/g, twice daily (Experimental): Participants applied 3 mcg/g CD2027 Ointment (up to 10 gram per application) topically, twice daily (at least 8 hours apart) over 4 weeks on atopic dermatitis lesions.
  Interventions: Drug: CD2027 Ointment 3 mcg/g, twice daily
- Vehicle Ointment, twice daily (Placebo Comparator): Participants applied Vehicle Ointment (up to 10 gram per application) topically, twice daily (at least 8 hours apart) over 4 weeks on atopic dermatitis lesions.
  Interventions: Drug: Vehicle Ointment, twice daily

INTERVENTIONS:
Drug: CD2027 Ointment 3 mcg/g, twice daily — Topical Ointment
  Arms: CD2027 Ointment 3 mcg/g, twice daily
Drug: Vehicle Ointment, twice daily — Topical Ointment
  Arms: Vehicle Ointment, twice daily

SUMMARY:
This was a multi-center, randomized, double-blind, parallel group study. Efficacy Objectives: To evaluate the efficacy of CD2027 ointment 3 mcg/g applied twice daily over 4 weeks versus its vehicle in adult participants with at least moderate atopic dermatitis.

Safety objective: To evaluate safety of CD2027 ointment 3 mcg/g when applied twice daily over 4 weeks versus its vehicle on 5 percent (%) - 20% involved Body Surface Area (BSA) (excluding Head/Neck) in adult participants with at least moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant, 18 years of age or older
* Clinical diagnosis of atopic dermatitis according to Hanifin and Rajka criteria, of at least moderate intensity according to Investigator Global Assessment (IGA greater or equal to 3)
* Body surface affected by the disease between 5% and 20% of total BSA, based on Rule of Nine's, excluding Head/Neck
* At least one area (Target Lesion) which was representative of the participant's disease state, was not located on the hands, feet or genitalia, measures at least 10 cm^2, presented a Total Severity Score of at least 6/15 (total severity score defined as the sum of Erythema, Excoriation, Papulation/Induration, Oozing/Crusting and Lichenification) with oozing/crusting severity at most 1

Exclusion Criteria:

* The participant had albumin-adjusted calcium above the upper normal range from screening evaluation
* The participant had history/signs/symptoms suggestive of an abnormality of calcium homeostasis (such as hyperparathyroidism, Paget's disease, adrenal insufficiency, hyperthyroidism)
* The participant had signs/symptoms of urinary stones or has a history of urinary stones within the past 5 years prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-05-21 (Actual); Primary Completion 2009-10-01 (Actual); Study Completion 2009-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (14):
- United States (14):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Therapeutics Clinical Research, Inc., San Diego, California
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - International Dermatology Research, Inc., Miami, Florida
  - Dermatology Specialists PSC, Louisville, Kentucky
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Helendale Dermatology & Medical Spa, LLC, Rochester, New York
  - Oregon Dermatology & Research Center, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Arlington Research Center, Inc., Arlington, Texas
  - DermResearch Inc., Austin, Texas
  - J&S Studies, Inc., College Station, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in the United States from 21 May 2009 to 01 October 2009.
Pre-assignment Details: A total of 147 participants were screened, of which 102 participants were enrolled and randomized to receive study treatment and 45 participants were reported as screen failure.
Groups:
- CD2027 Ointment 3 mcg/g, Twice Daily: Participants applied 3 microgram per gram (mcg/g) CD2027 Ointment (up to 10 gram per application) topically, twice daily (at least 8 hours apart) over 4 weeks on atopic dermatitis lesions.
Period: Overall Study
Arm/Group | CD2027 Ointment 3 mcg/g, Twice Daily | Vehicle Ointment, Twice Daily
Started | 53 | 49
Completed | 41 | 45
Not Completed | 12 | 4
Not completed — Adverse Event | 7 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed on Intent To Treat (ITT) Population that included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CD2027 Ointment 3 mcg/g, Twice Daily | Vehicle Ointment, Twice Daily | Total
Number analyzed (Participants) | 53 | 49 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 48 | 98
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (14.9) | 40.3 (13.8) | 39.3 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 20 | 48
  Male | 25 | 29 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4 | 5 | 9
  Race: Black | 5 | 10 | 15
  Race: Caucasian | 27 | 21 | 48
  Race: Hispanic | 15 | 10 | 25
  Race: OTHER | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 49 | 102

OUTCOME MEASURES:

1. Primary Outcome: Total Severity Score (TSS) of Target Lesion at Baseline and Week 4
Description: TSS comprised of the sum of an assessment of erythema, excoriation, exudation, lichenification and pruritus, each on a scale of 0 to 3 to give a maximum score of 15; 0 (best) and 3 (worst) indicated total possible minimum score was 0 and total possible maximum score was 15. Lower score meant improvement in condition and higher score indicated worsening of condition.
Time Frame: Baseline, Week 4
Population: Intent To Treat (ITT) Population included all randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD2027 Ointment 3 mcg/g, Twice Daily | Vehicle Ointment, Twice Daily
Number analyzed (Participants) | 53 | 49
score on a scale
  Baseline | 7.62 (1.47) | 7.49 (1.53)
  Week 4 | 4.7 (2.6) | 4.6 (3.2)

2. Secondary Outcome: Change From Baseline in Total Severity Score (TSS) for Individual Signs at Week 4
Description: TSS comprised of the sum of an assessment of erythema, excoriation, exudation, lichenification and pruritus, each on a scale of 0 to 3 to give a maximum score of 15; 0 (best) and 3 (Worst) indicated total possible minimum score was 0 and total possible maximum score was 15. Data for individual signs is reported in this outcome measure. Lower score meant improvement in condition and higher score indicated severity (worsening of condition) for each individual sign.
  Erythema was evaluated on a four point scale of 0 to 3 where (0=none, 1=mild, 2=moderate, 3=severe). Excoriation evaluated on a four point scale of 0 to 3 where (0=none, 1=mild, 2=moderate, 3=severe). Exudation was evaluated on a four point scale of 0 to 3 where (0=none, 1=mild, 2=moderate, 3=severe). Lichenification was evaluated on a four point scale of 0 to 3 where (0=none, 1=mild, 2=moderate, 3=severe). Pruritus was evaluated on a four point scale of 0 to 3 where (0=none, 1=mild, 2=moderate, 3=severe).
Time Frame: Baseline, Week 4
Population: ITT Population included all randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD2027 Ointment 3 mcg/g, Twice Daily | Vehicle Ointment, Twice Daily
Number analyzed (Participants) | 53 | 49
score on a scale
  Erythema | -0.7 (0.9) | -0.7 (0.7)
  Induration/Papulation | -0.7 (0.9) | -0.7 (0.8)
  Excoriation | -0.8 (0.9) | -0.7 (0.7)
  Lichenification | -0.5 (0.7) | -0.6 (0.8)
  Pruritus | -0.9 (1.1) | -0.8 (1.2)

3. Secondary Outcome: Number of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" and Failure From Baseline of Greater Than 1 Points Over Week 4
Description: IGA was an assessment scale used to determine severity of Atopic Dermatitis (AD) and clinical response to treatment on a 5-point scale (0=clear; 1=almost clear; 2=mild; 3=moderate; 4=severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score of "0" or "1" and a failure from baseline of greater than (>1) points over 4 weeks were reported.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: ITT Population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CD2027 Ointment 3 mcg/g, Twice Daily | Vehicle Ointment, Twice Daily
Number analyzed (Participants) | 53 | 49
Participants
  Baseline: Success (IGA=0 or 1) | 0 | 0
  Baseline: Failure (IGA>1) | 53 | 49
  Week 1: Success (IGA=0 or 1) | 2 | 0
  Week 1: Failure (IGA>1) | 51 | 49
  Week 2: Success (IGA=0 or 1) | 3 | 1
  Week 2: Failure (IGA>1) | 50 | 48
  Week 3: Success (IGA=0 or 1) | 5 | 3
  Week 3: Failure (IGA>1) | 48 | 46
  Week 4: Success (IGA=0 or 1) | 10 | 11
  Week 4: Failure (IGA>1) | 43 | 38

4. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 1, 2, 3, 4
Description: The EASI score quantifies the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on a scale of 0 (none) to 3 (severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions was scored on a scale of 0 (no eruption) to 6 (>90%-100% eruption). The total score was the sum of the four body-region scores, maximum=72, minimum=0, Higher scores indicated greater disease severity.
Time Frame: Baseline, Week1, Week2, Week 3, Week 4
Population: ITT Population included all randomized participants.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CD2027 Ointment 3 mcg/g, Twice Daily | Vehicle Ointment, Twice Daily
Number analyzed (Participants) | 53 | 49
percent change
  Week 1 | -10.0 (34.2) | -16.2 (34.2)
  Week 2 | -21.3 (51.3) | -26.7 (36.9)
  Week 3 | -28.7 (63.3) | -33.2 (41.6)
  Week 4 | -29.6 (69.9) | -41.4 (45.7)

ADVERSE EVENTS:
Time Frame: Up to 4 months.
Description: Safety analysis set included all randomized participants who applied the study medication.
Arm/Group | CD2027 Ointment 3 mcg/g, Twice Daily | Vehicle Ointment, Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/49
Other Adverse Events (participants affected / at risk) | 16/53 | 8/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD2027 Ointment 3 mcg/g, Twice Daily (N=53) | Vehicle Ointment, Twice Daily (N=49)
Application site pruritis (General disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Blood 1,25-dihydroxycholecalciferol increased (Investigations) | 5 (5) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes